CLINICAL TRIAL: NCT06251232
Title: Proof-of-concept Phase II Study to Evaluate the Efficacy and Safety of Prednisone in the Treatment of Idiosyncratic Hepatotoxicity and Its Mechanistic Pathways Through an Integrative Analysis: the DILI-CORT Clinical Trial
Brief Title: Proof-of-concept to Evaluate the Efficacy and Safety of Prednisone in Idiosyncratic Hepatotoxicity
Acronym: DILICORT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DILICORT
Record Dates: First submitted 2023-12-12; First posted 2024-02-09 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-11

CONDITIONS: Hepatotoxicity; Idiosyncratic Drug Effect; Prednisone
Keywords: Prednisone; Idiosyncrasic hepatotoxicity
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Controlled with placebo
Who Masked: Outcomes Assessor
Masking Description: Prednisone medication and its placebo will be identical in appearance and in organoleptic properties.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Active Comparator): Oral prednisone
  Interventions: Drug: Prednisone
- Placebo treatment (Placebo Comparator): Placebo
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Placebo
  Other Names: Comparator

SUMMARY:
This trial´s aim is to assess if oral prednisone (compared to placebo), administered over five weeks is beneficial in terms of decreased total bilirubin (TBL): reduction of the peak of TBL at least 50% at 14 days or reduction in the time to normalisation of TBL value.

DETAILED DESCRIPTION:
This trial´s aim is to assess if oral prednisone (compared to placebo), administered over five weeks is beneficial in terms of decreased total bilirubin (TBL): reduction of the peak of TBL at least 50% at 14 days or reduction in the time to normalisation of TBL value, and to assess if oral prednisone (compared to placebo) is safe and well tolerated in patients with acute moderate to severe DILI.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients, aged ≥ 18 years.
2. Patients who have been diagnosed with DILI by the expert committee.
3. Patients with moderate to severe DILI (elevations of ALT or AST ≥ 5 times the Upper Limit of Normal (ULN) and serum TBL ≥ 2.5 mg/dL).
4. Patients who do not show a 15% reduction in ALT values or TBL continues to increase 5-10 days after liver damage recognition despite the withdrawal of the culprit drug.

Exclusion Criteria:

1. No clear DILI diagnosis after an expert committee DILI assessment.
2. DILI due to immune-checkpoint inhibitors.
3. Presence of active infection as evidenced by positive urine or blood culture.
4. Acute liver failure (international normalized ratio (INR) > 1.5 and hepatic encephalopathy).
5. Model for End-Stage Liver Disease (MELD) ≥ 30.
6. Known hypersensitivity to prednisone or placebo components.
7. Pregnant or nursing mothers.
8. Co-existing infection with hepatitis C, hepatitis B, or human immunodeficiency virus (HIV).
9. Patients already receiving systemic steroids or other immunosuppressants.
10. Inability to provide informed consent.
11. Presence of clinically significant comorbid illnesses (by clinician's criteria) that might impede the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Total bilirubin | Through study completation, an average 2 years
  To assess if oral prednisone (compared to placebo), administered over five weeks is beneficial in terms of decreased total bilirubin (TBL): reduction of the peak of TBL at least 50% at 14 days or reduction in the time to normalisation of TBL value.

SECONDARY OUTCOMES:
Peak alanine aminotransferase level | 2 years
  Comparison prednisone/placebo when reducing peak alanine aminotransferase (ALT), aspartate aminotransferase (AST) and international normalized ratio (INR) values by at least 50% at day 7 or reducing the time to normalisation.
Aspartate aminotransferase level | 2 years
  Comparison prednisone/placebo when reducing peak alanine aminotransferase (ALT), aspartate aminotransferase (AST) and international normalized ratio (INR) values by at least 50% at day 7 or reducing the time to normalisation.
International normalized ratio values | Through study completation, an average 2 years
  Comparison prednisone/placebo when reducing peak alanine aminotransferase (ALT), aspartate aminotransferase (AST) and international normalized ratio (INR) values by at least 50% at day 7 or reducing the time to normalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Raúl Andrade, PhD, Principal Investigator — SAS

IPD SHARING:
Plan to Share IPD: Yes
National and international webs, manuscript
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After 3 years
Access Criteria: Open access